CLINICAL TRIAL: NCT04006639
Title: Comparison of Efficacy Between Bilateral Superficial Cervical Plexus Block and Local Infiltration of Lidocaine 2% in Patients Undergoing Tracheostomy
Brief Title: Efficacy of Bilateral Superficial Cervical Plexus Block vs. Local Infiltration of Lidocaine 2% in Tracheostomy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pryambodho Pryambodho, Medical Staff in Department of Anesthesiology and Intensive Care, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes029
Record Dates: First submitted 2019-05-27; First posted 2019-07-05 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Tracheostomy
Keywords: local infiltration; bilateral superficial cervical plexus block; lidocaine; bupivacaine; substance-p

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral superficial cervical plexus block with Bupiv (Active Comparator): Patients, who will have tracheostomy procedure, might receive bilateral superficial cervical plexus block with 10 mL of Bupivacaine 0.5% (20 mL spuit with 25 G 1.5 inch needle) on each side before tracheostomy procedure.
  Interventions: Procedure: Analgesic Technique
- Local infiltration of Lidocaine 2% (Active Comparator): Patients, who will have tracheostomy procedure, might receive local infiltration of Lidocaine 2% (5 mL spuit with 25 G 1.5 inch needle) before tracheostomy procedure.
  Interventions: Procedure: Analgesic Technique

INTERVENTIONS:
Procedure: Analgesic Technique — Patients undergoing tracheostomy procedure must be administered with analgesics, such Lidocaine 20% or Bupivacaine 0.5%

SUMMARY:
The aim of this study was to compare the efficacy between superficial cervical plexus block and local infiltration of lidocaine 2% in patients undergoing tracheostomy procedure.

DETAILED DESCRIPTION:
Ethical approval was obtained from Ethics Committee of Faculty of Medicine, Universitas Indonesia - Dr. Cipto Mangunkusumo Hospital.

Eligible subjects for this study will be recruited with consecutive sampling method within certain period until minimum number of subjects required for this study is filled.

Informed consents will be given to each subject before participating in the study. Patients will be randomly divided into two groups using closed envelops.

Subjects who will receive bilateral superficial cervical plexus block is the interventional group whereas subjects who will receive local infiltration of lidocaine 2% is the control group.

Before, during, and after the procedure, all subjects are monitored (blood pressure, heart rate, respiratory rate, and electrocardiography). Monitoring data, including pain, will be recorded. Pain is measured by using visual analog scale or verbal numeric rating scale.

Arterial blood sample (approximately 3 cc) from each subject will be withdrawn twice and put into tubes containing anticoagulant for substance-P examination. Initial withdrawal is done before the anesthetics are given while the last one is done after the tracheostomy procedure.

Before the procedure, location for incision and block will be marked. Interventional group will be given 10 mL of Bupivacaine 0.5% on each side of the neck (as marked) by using 20 mL spuit with 25 G 1.5 inch needle whereas control group will be given 4 mL of Lidocaine 2% on incisional region (as marked) by using 5 mL spuit with 25 G 1.5 inch needle. 1 mg of Midazolam can be given intravenously before the block if there is no contraindication. Tracheostomy will be performed 15 minutes after the block is administered or local infiltration has worked. After tracheostomy, patients will be continually monitored in post-anesthesia care unit while their blood samples will be delivered to laboratory for ELISA test.

ELIGIBILITY:
Inclusion Criteria:

* Physical Status ASA 1-3

Exclusion Criteria:

* Pregnant
* Blood clotting disorder
* Allergic to anesthetics (Lidocaine, Bupivacaine) used in this study
* Local infection on procedure area
* Deformity on procedure area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Concentration of substance-P (Baseline) | 3 months
  Substance-P level is measured as a pain indicator.
Concentration of substance-P (After Tracheostomy) | 3 months
  Substance-P level is measured as a pain indicator.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pandit JJ, Satya-Krishna R, Gration P. Superficial or deep cervical plexus block for carotid endarterectomy: a systematic review of complications. Br J Anaesth. 2007 Aug;99(2):159-69. doi: 10.1093/bja/aem160. Epub 2007 Jun 18. PMID 17576970
- [Result] Brandow AM, Wandersee NJ, Dasgupta M, Hoffmann RG, Hillery CA, Stucky CL, Panepinto JA. Substance P is increased in patients with sickle cell disease and associated with haemolysis and hydroxycarbamide use. Br J Haematol. 2016 Oct;175(2):237-245. doi: 10.1111/bjh.14300. Epub 2016 Aug 19. PMID 27539682
- [Result] Douglas SD. Substance P and sickle cell disease-a marker for pain and novel therapeutic approaches. Br J Haematol. 2016 Oct;175(2):187-188. doi: 10.1111/bjh.14299. Epub 2016 Aug 19. No abstract available. PMID 27539537
- [Result] De Leyn P, Bedert L, Delcroix M, Depuydt P, Lauwers G, Sokolov Y, Van Meerhaeghe A, Van Schil P; Belgian Association of Pneumology and Belgian Association of Cardiothoracic Surgery. Tracheotomy: clinical review and guidelines. Eur J Cardiothorac Surg. 2007 Sep;32(3):412-21. doi: 10.1016/j.ejcts.2007.05.018. Epub 2007 Jun 27. PMID 17588767
- [Result] Fernandez-Bussy S, Mahajan B, Folch E, Caviedes I, Guerrero J, Majid A. Tracheostomy Tube Placement: Early and Late Complications. J Bronchology Interv Pulmonol. 2015 Oct;22(4):357-64. doi: 10.1097/LBR.0000000000000177. PMID 26348694
- [Result] Griffiths J, Barber VS, Morgan L, Young JD. Systematic review and meta-analysis of studies of the timing of tracheostomy in adult patients undergoing artificial ventilation. BMJ. 2005 May 28;330(7502):1243. doi: 10.1136/bmj.38467.485671.E0. Epub 2005 May 18. PMID 15901643
- [Result] Mehta C, Mehta Y. Percutaneous tracheostomy. Ann Card Anaesth. 2017 Jan;20(Supplement):S19-S25. doi: 10.4103/0971-9784.197793. PMID 28074819